CLINICAL TRIAL: NCT07275645
Title: A Phase III, Randomized, Blinded, and Homologous Vaccine-Controlled Clinical Trial to Evaluate the Immunogenicity and Safety of the Rabies Vaccine (Human Diploid Cell), Freeze-dried, Vaccinated With Different Immunization Schedules in a Population Aged 10 to 60 Years
Brief Title: A Clinical Trial of Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried in a Population Aged 10 to 60 Years
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ab&B Bio-tech Co., Ltd.JS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HDCV-ZHSW-04
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Rabies
Keywords: Rabies; Rabies vaccine
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Essen Control Group (Active Comparator)
  Interventions: Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried
- Essen Experimental Group (Experimental)
  Interventions: Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried
- Zagreb Experimental Group (Experimental)
  Interventions: Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried
- Simplified Four-Dose Group 1 (Experimental)
  Interventions: Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried
- Simplified Four-Dose Group 2 (Experimental)
  Interventions: Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried

INTERVENTIONS:
Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried — The vaccine will be administered via intramuscular injection into the deltoid muscle of the upper arm, with a human dose of 1.0 ml per injection. A total of 5 doses will be administered at Day 0, 3, 7, 14, and 28. Some participants will also undergo re-exposure immunization, receiving one additional dose of the vaccine on Days 0 and 3 of the re-exposure phase.
  Arms: Essen Experimental Group
Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried — The vaccine will be administered via intramuscular injection into the deltoid muscle of the upper arm, with a human dose of 1.0 ml per injection. Two doses will be administered on Day 0, followed by one dose each on Days 7 and 21, for a total of 4 doses. Some participants will also undergo re-exposure immunization, receiving one additional dose of the vaccine on Days 0 and 3 of the re-exposure phase.
  Arms: Zagreb Experimental Group
Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried — The vaccine will be administered via intramuscular injection into the deltoid muscle of the upper arm, with a human dose of 1.0 ml per injection. A total of 4 doses will be administered at Day 0, 3, 7 and 14. Some participants will also undergo re-exposure immunization, receiving one additional dose of the vaccine on Days 0 and 3 of the re-exposure phase.
  Arms: Simplified Four-Dose Group 1
Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried — The vaccine will be administered via intramuscular injection into the deltoid muscle of the upper arm, with a human dose of 1.0 ml per injection. A total of 4 doses will be administered at Day 0, 3, 7, and 28. Some participants will also undergo re-exposure immunization, receiving one additional dose of the vaccine on Days 0 and 3 of the re-exposure phase.
  Arms: Simplified Four-Dose Group 2
Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried — The vaccine will be administered via intramuscular injection into the deltoid muscle of the upper arm, with a human dose of 1.0 ml per injection. A total of 5 doses will be administered at Day 0, 3, 7, 14, and 28.
  Arms: Essen Control Group

SUMMARY:
A total of 3,000 participants will be enrolled, stratified by age into two groups: 600 participants aged 10-17 years and 2,400 participants aged 18-60 years. Within each age group, participants will be randomly assigned in a 1:1:1:1:1 ratio to one of five vaccination schedule groups: Essen Control Group (Group A), Essen Experimental Group (Group B), Zagreb Experimental Group (Group C), Simplified Four-Dose Group 1 (Group D), and Simplified Four-Dose Group 2 (Group E).

Among participants in the four experimental groups-Essen Experimental Group, Zagreb Experimental Group, Simplified Four-Dose Group 1, and Simplified Four-Dose Group 2-stratified block randomization will be applied. Within each age group and each vaccination schedule group, participants will be further randomized in a 1:1:1 ratio into three subgroups: those receiving a booster dose at Day 90 after completion of the primary immunization, those receiving a booster dose at Day 180, and those undergoing assessment of immune persistence at Day 360 after completion of the primary immunization.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 10 and 60 years at the time of enrollment.
* The participant and/or their legal guardian voluntarily agrees to participate in the trial and signs the informed consent form.
* The participant and their family are able to comply with the trial follow-up schedule as required by the protocol (no plans for extended absence or relocation from the study site).
* Female participants are neither pregnant nor lactating (negative urine pregnancy test prior to vaccination), and have no plans to become pregnant within 2 months after enrollment.

Exclusion Criteria:

a Exclusion criteria for the first dose:

* Axillary body temperature ≥37.3°C at screening.
* History of rabies vaccination or administration of rabies-specific passive immunization products, or history of bites/scratches by dogs or other mammals within the past year.
* History of severe allergic reactions requiring medical intervention to any vaccine or vaccine components, such as anaphylactic shock, allergic laryngeal edema, allergic purpura, Arthus reaction, severe urticaria, or angioedema.
* Fever, acute or chronic infectious diseases (e.g., active tuberculosis, viral hepatitis), or acute exacerbation of chronic illness within 3 days before the first vaccine dose.
* Receipt of blood, blood products, or immunoglobulins within 3 months prior to the first vaccine dose, or planned use of such products within 1 month after the final vaccine dose.
* Receipt of any other vaccines within 14 days prior to the first vaccine dose.
* Asplenia or functional asplenia due to any condition (e.g., splenectomy).
* Diagnosed congenital or acquired immunodeficiency (including HIV infection), or treatment with immunosuppressive agents within the past 3 months (e.g., systemic corticosteroids for ≥14 days at doses ≥2 mg/kg/day or ≥20 mg/day of prednisone or equivalent).
* Presence of severe congenital malformations, autoimmune (hereditary) diseases, or severe chronic conditions (including but not limited to: thalassemia, heart disease, kidney disease, diabetes, hereditary allergic constitution, Guillain-Barré syndrome, etc.)
* Personal or family history of convulsions, epilepsy, encephalopathy, or psychiatric disorders.
* Contraindications to intramuscular injection (e.g., diagnosed thrombocytopenia, any coagulation disorder, or current use of anticoagulant therapy).
* Uncontrolled hypertension (e.g., systolic BP ≥160 mmHg and/or diastolic BP ≥100 mmHg at screening for adults aged 18 years and above).
* Currently participating in another clinical trial involving investigational or unregistered products (drugs or vaccines), or planning to participate in another clinical trial before completion of this study.
* Any condition that, in the opinion of the investigator, may interfere with the evaluation of the study objectives.

b Exclusion criteria for subsequent doses:

* Positive urine pregnancy test；
* Severe anaphylaxis after the previous dose;
* Grade 4 adverse events associated with trial vaccination after the previous dose;
* Exposure during the course (bite or scratch from dogs, cats or other mammals);
* Participant has any other conditions that warrant discontinuation of vaccination as determined by the investigator.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-12-18 (Estimated); Primary Completion 2026-02-18 (Estimated); Study Completion 2027-02-18 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate and geometric mean concentration (GMC) of rabies virus neutralizing antibodies in baseline seronegative participants 14 days after the first dose. | Day 14 after the first dose.
Seroconversion rate of rabies virus neutralizing antibodies in baseline seronegative participants 14 days after the last dose. | Day 14 after the last dose.
Incidence of adverse events within different timeframes (30 minutes, 0-7 days, 0-30 days) after each vaccine dose. | Within 30 minutes, 0-7 days, and 0-30 days after each dose
All serious adverse events (SAEs) occurring from the first dose of primary immunization to 6 months after completion of the primary immunization. | From the first dose of primary immunization to 6 months after completion

SECONDARY OUTCOMES:
Geometric mean concentration (GMC) of rabies virus neutralizing antibodies in baseline seronegative participants 14 days after the last dose. | Day 14 after the last dose
Comparison of seroconversion rates and GMCs among baseline seronegative participants in the Essen Experimental Group, Simplified Four-Dose Group 1, and Simplified Four-Dose Group 2 at Days 28 and 42 after the first dose. | Days 28 and 42 after the first dose
Comparison of seroconversion rates and GMCs in baseline seronegative participants between the Essen Experimental Group and the Zagreb Experimental Group at Day 7 after the first dose. | Day 7 after the first dose

OTHER OUTCOMES:
Seropositivity rate and GMC of rabies virus neutralizing antibodies in a subset of participants at 90 days, 180 days, and 360 days after completion of the primary immunization. | 90, 180, and 360 days post-primary immunization
Seropositivity rate and GMC in a subset of participants at 14, 42, 90, and 180 days after the first dose of re-exposure immunization. | 14, 42, 90, and 180 days after re-exposure immunization

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Qichun County Center for Disease Control and Prevention, Huanggang, Hubei
  - Yunyang District Center for Disease Control and Prevention, Shiyan, Hubei
  - Zhushan county Center for Disease control and Prevention, Shiyan, Hubei
  - Gucheng county Center for Disease control and Prevention, Xiangyang, Hubei
  - Xiangzhou District Center for Disease Control and Prevention, Xiangyang, Hubei

IPD SHARING:
Plan to Share IPD: No